CLINICAL TRIAL: NCT02335346
Title: An Open Label Extension Study of Phase 3 Trial of Duloxetine in Patients With Osteoarthritis and Knee Pain
Brief Title: An Extension Study of Duloxetine in Osteoarthritis and Knee Pain (Extension of F1J-JE-HMGX, NCT02248480)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15611; F1J-JE-HMHD (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental): Duloxetine 20 milligram (mg) for first week, 40 mg for second week and 60 mg for next 48 weeks administered orally once daily. During tapering period, dose of 40 mg for one week and then 20 mg for the last week.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: LY248686; Cymbalta

SUMMARY:
The purpose of this study is to assess the safety and efficacy of duloxetine in participants with osteoarthritis and knee pain. The study will last for 1 year.

ELIGIBILITY:
Inclusion Criteria:

(Consecutive Participants)

* Participants who have completed the 15-week treatment in the preceding study HMGX.

(New Participants)

* Participants with present osteoarthritis (OA) based on American College of Rheumatology (ACR) classification of idiopathic OA of the knee.
* Have pain for ≥14 days of each month for 3 months prior to study entry.
* Have a score of ≥4 on the BPI average pain score at the start of the study.

(Consecutive and New Participants)

* Females of child-bearing potential must test negative (-) on a pregnancy test.

Exclusion Criteria:

(New Participants)

* Participants who have any previous diagnosis of psychosis, bipolar disorder, or schizoaffective disorder.
* Participants who have major depressive disorder as determined using depression module of the Mini-International Neuropsychiatric Interview (M.I.N.I.).
* Participants who have received intrarticular hyaluronate or steroids, joint lavage, or other invasive therapies to the knee in the past 1 week.
* Participants who have had knee arthroscopy of the index knee within the past year or joint replacement of the index knee or osteotomy at any time.
* Participants have a prior synovial fluid analysis showing a white blood cell (WBC) ≥2000 cubic millimeters (mm3) that is indicative of a diagnosis other than OA.
* Participants who have a history of having more than one medical allergy.
* Are non-ambulatory or require the use of crutches or a walker.
* Have frequent falls that could result in hospitalization or could compromise response to treatment.
* Have a history of drug abuse or dependence within the past year, including alcohol and excluding nicotine and caffeine.
* Have a positive urine drug screen for any substances of abuse or excluded medication.
* Have received administration of another investigational drug within the 30 days prior to enrollment.
* Have had previous exposure to duloxetine or completed/withdrawn from any study investigating duloxetine.

(Consecutive and New Participants)

* Participants who have serious cardiovascular, hepatic, renal, endocrine, respiratory, or hematologic illness, peripheral vascular disease, or other medical condition or neuropsychiatric conditions or clinically significant laboratory abnormalities or electrocardiographic abnormalities.
* Participants who have alanine aminotransferase (ALT) or aspartate aminotransferase (AST) higher than 100 international units per liter (IU/L) or total bilirubin higher than 1.6 milligrams/deciliter (mg/dL).
* Participants having serum creatinine level higher than 2.0 mg/dL, or had renal transplantation or receiving renal dialysis.
* Participants who have a diagnosis of inflammatory arthritis (that is, rheumatoid arthritis) or an autoimmune disorder (excluding inactive Hashimoto's thyroiditis and Type 1 diabetes).
* Participants who have uncorrected thyroid disease, uncontrolled narrow-angle glaucoma, history of uncontrolled seizures, or uncontrolled or poorly controlled hypertension.
* Participants who have end stage bone disease or surgery planned during the trial for the index joint.
* Participants treated with a monoamine oxidase inhibitor (MAO) within 14 days prior to baseline, or those with the potential need to use MAO inhibitor during the study or within 5 days of discontinuation of investigational drug.
* Participants who answer 'yes' to any of the questions about active suicidal ideation/intent/behaviors occurring within the past month (Columbia-Suicide Severity Rating Scale, suicide ideation section-questions 4 and 5; suicidal behaviors section).
* Have a primary painful condition that may interfere with assessment of the index joint, i.e., knee.
* Pregnant participants, female participants who wish to be pregnant during the clinical study period, or participants who are breast-feeding; or male participants who wish pregnancy of the partner.
* Participants who cannot use appropriate contraceptive method or do not want to use that from the start of the study until one month after the end of administration of the investigational drug.
* Considered as inappropriate participation to the study for any medical or other reason by the investigator.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kobe, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were consecutive participants from F1J-JE-HMGX, NCT02248480. No new participants were enrolled.
Period: Overall Study
Arm/Group | Duloxetine
Started | 93
Received At Least 1 Dose of Study Drug | 93
Completed | 81
Not Completed | 12
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Duloxetine: Duloxetine 20 mg for first week, 40 mg for second week and 60 mg for next 48 weeks administered orally once daily. During tapering period, dose of 40 mg for one week and then 20 mg for the last week.
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 93
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug Related Adverse Events (AEs) or Any Serious Adverse Events (SAEs)
Description: A summary of drug related (considered by the investigator) AEs and SAEs is located in the Reported Adverse Events module. An AE is summarized if the onset date is on or after the first dose of study drug and within 7 days after the last dose, or it occurred before the first dose of study drug and worsened while on the therapy.
Time Frame: Baseline through Week 53
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
Percentage of participants
  Drug-Related Adverse Event | 51.6
  Serious Adverse Event | 7.5

2. Secondary Outcome: Patient Global Impression-Improvement (PGI-I) at 50 Weeks
Description: Patient Global Impressions of Improvement Scale: PGI-I measures a participant's perception of improvement at the time of assessment compared with the start of treatment. Score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Week 50
Population: All enrolled participants who received at least one dose of study drug. Missing values due to discontinuation of study or drug, or missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
units on a scale | 2.09 (0.94)

3. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) to Week 50
Description: CSI-S measures severity of illness at the time of assessment compared with start of treatment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline, Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
units on a scale | -2.19 (0.99)

4. Secondary Outcome: Change From Baseline to 50 Weeks on the Brief Pain Inventory-Severity and Interference Rating Short Form (BPI-SF)
Description: Brief Pain Inventory Severity and Interference Scores: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items.
Time Frame: Baseline, Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
units on a scale
  Worst Pain | -4.29 (2.05)
  Least Pain | -2.16 (1.66)
  Average Pain | -3.33 (1.81)
  Pain Right Now | -2.94 (2.19)
  General Activity | -3.03 (2.22)
  Mood | -2.48 (2.25)
  Walking Ability | -3.11 (2.17)
  Normal Work | -3.10 (2.41)
  Relationship People | -1.43 (2.07)
  Sleep | -1.81 (2.35)
  Enjoy of Life | -1.92 (2.16)
  Average of 7 items | -2.41 (1.81)

5. Secondary Outcome: Change From Baseline to 50 Weeks on the Western Ontario and McMaster Osteoarthritis Index (WOMAC) Questionnaire Total Score
Description: The 24-question WOMAC Osteoarthritis Index assesses osteoarthritis symptoms using pain (5 questions), stiffness (2 questions) and physical function (17 questions) subscales. The WOMAC Osteoarthritis Index version 3.1 was administered according to the study schedule. The WOMAC total score was calculated for each participant at each time point for analysis as the mean total score, range 0 (none) -96 millimeter (mm)(extreme).
Time Frame: Baseline, Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
units on a scale | -20.23 (15.05)

6. Secondary Outcome: Change From Baseline to 50 Weeks on the 36-Item Short-Form Health Survey (SF-36)
Description: 36-item Short-Form Health Survey: SF-36 Health Status Survey is a generic, health-related scale assessing participant's quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. Domain scores: general health (range: 5-25); physical functioning (range: 10-30); role-physical (range: 4-8); role-emotional (range: 3-6); social functioning (range: 2-10); bodily pain (range: 2-11); vitality (range: 4-24); mental health (range: 5-30).
Time Frame: Baseline, Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
units on a scale
  Physical Functioning | 15.27 (20.82)
  Role (Physical) | 11.90 (21.20)
  Bodily Pain | 21.32 (21.15)
  General Health | 10.89 (17.20)
  Vitality | 9.61 (16.16)
  Social Functioning | 6.45 (19.12)
  Role(Emotional) | 8.78 (23.13)
  Mental Health | 4.89 (18.37)

7. Secondary Outcome: Change From Baseline to 50 Weeks on the 5 Dimension (EQ-5D) Version of the European Quality of Life Instrument
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument.The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a three level scale (no problem, some problems, and major problems). These combinations of attributes were converted into a weighted health-state Index Score according to the Japan population-based algorithm with scores ranging from -0.111 to 1.0. A higher score indicates better health state.
Time Frame: Baseline, Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
units on a scale | 0.15 (0.16)

8. Secondary Outcome: Change From Baseline to 50 Weeks on the Beck Depression Inventory (BDI-II) Total Score
Description: Beck Depression Inventory-II: BDI-II is a 21-item, participant-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to symptoms of depression were scored on a 4-point scale ranging from 0 to 3 and was summed to give a single score. A total score of 0-13 was considered minimal range, 14-19 was mild, 20-28 was moderate, and 29-63 was severe.
Time Frame: Baseline, Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
units on a scale | -1.14 (4.93)

9. Secondary Outcome: Percentage of Participants With Fall Events From Fall Questionnaire
Description: Participants reported the details of their falls. Percentage equals the number of participants with fall events / total in treatment group * 100.
Time Frame: Baseline through Week 50
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 93
Percentage of Participants | 23.7

ADVERSE EVENTS:
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 7/93
Other Adverse Events (participants affected / at risk) | 85/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=93)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Progressive supranuclear palsy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine (N=93)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Chalazion (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 18 (20)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 2 (2)
Thirst (General disorders) | 11 (11)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 5 (6)
Chronic sinusitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 2 (3)
Gastroenteritis (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (21)
Onychomycosis (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 3 (3)
Otitis media chronic (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (2)
Pharyngitis (Infections and infestations) | 4 (4)
Purulence (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Tinea pedis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (3)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 8 (11)
Epicondylitis (Injury, poisoning and procedural complications) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Frostbite (Injury, poisoning and procedural complications) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 6 (6)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Urobilinogen urine increased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myofascitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Intercostal neuralgia (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 3 (3)
Somnolence (Nervous system disorders) | 12 (12)
Disorientation (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Neurosis (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (2)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/26 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Yellow skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 7 (7)
Lymphoedema (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days